CLINICAL TRIAL: NCT04697901
Title: Sustaining Aviator Performance During Extended Operational Flight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Aeromedical Research Laboratory (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: USAARL 2019-014; IRB M-10804
Record Dates: First submitted 2020-06-08; First posted 2021-01-06 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Stimulation (Experimental): Active tDCS stimulation will be applied.
  Interventions: Device: Active Transcranial Direct Current Stimulation (tDCS)
- Sham Stimulation (Sham Comparator): Sham tDCS stimulation will be applied.
  Interventions: Device: Sham Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Active Transcranial Direct Current Stimulation (tDCS) — Active simulation will be applied to the right PPC. To target this region for stimulation, the anode electrode will be placed on the subject using the 10-20 EEG system as reference location (Thair et al., 2017). Stimulation intensity for all conditions will be set to 2 mA, which was chosen based on previous studies that have compared 1 mA to 2 mA and found the higher intensity produced reliable changes to performance (e.g., Moos et al., 2012). Total time of active stimulation will be the same for each group (20 minutes). Delivery times of the stimulation will vary based on Group assignment:
  Group A: During pre-flight brief/checklist, for 20 minutes. Group B: First delivered at 30 minutes into flight for 10 minutes, second delivered at 60 minutes into flight for 10 minutes.
  Arms: Active Stimulation
Device: Sham Transcranial Direct Current Stimulation (tDCS) — Sham simulation will be applied to the right PPC. To target this region for stimulation, the anode electrode will be placed on the subject using the 10-20 EEG system as reference location (Thair et al., 2017). Stimulation intensity for all conditions will be set to 2 mA, which was chosen based on previous studies that have compared 1 mA to 2 mA and found the higher intensity produced reliable changes to performance (e.g., Moos et al., 2012). Total time of active stimulation will be the same for each group (20 minutes). Sham stimulation will consist of active stimulation for 120s, including the ramping up to 2 mA and down to no stimulation. Delivery times of the stimulation will vary based on Group assignment:
  Group A: During pre-flight brief/checklist, for 20 minutes. Group B: First delivered at 30 minutes into flight for 10 minutes, second delivered at 60 minutes into flight for 10 minutes.
  Arms: Sham Stimulation

SUMMARY:
Future aviation operations are anticipated to change as advances in technology enable automation of more tasks. Development of new platforms under the Future Vertical Lift program are also anticipated to change the nature of missions as they are being designed to cover further distances. Longer duration flights coupled with greater automated features are expected to shift the role of the aviator, resulting in an increased need for attention maintenance, which creates potential problems related to performance. To offset the likelihood of performance decrements related to the need to sustain attention, we propose examining the use of transcranial electrical current stimulation. In the present study, we will evaluate whether delivery of stimulation prior to or during the task enables sustainment of attention and thereby reduces performance decrements as measured through primary flight tasks and a secondary attentional task. Further, we will evaluate whether stimulation enhances the ability to respond to an unexpected emergency toward the end of the flight.

DETAILED DESCRIPTION:
Volunteers will first schedule an appointment to complete informed consent, screening procedures and meet with study physician. After eligibility is verified, volunteers will complete baseline assessments. At the completion of baseline assessments volunteers will be scheduled for their return visits and will be given their actiwatch. Scheduling will occur such that there is at least 16 hours' time between baseline assessments and their first treatment visit, whereas treatment visits will be scheduled such that there is at least 48 hours between visits. Stimulation will be counterbalanced with at least 48 hours between deliveries to allow for a washout period (Nitsche & Paulus, 2001). Scheduling will be done such that individual participants are always scheduled at the same time of day to control for any effects of circadian rhythm and individual differences.

Visit 1: Test scheduling, informed consent, screening procedures and baseline assessments.

During this visit, subjects will be informed that they should have 8 hours of sleep the night before each testing session, with a minimum of 6 accepted for participation (confirmed by an actiwatch and self-report). A minimum of 6 hours will be accepted to avoid potential loss of subjects who are not able to obtain 8 hours. However, 8 hours will be stressed to encourage subjects to be well rested prior to the testing days. They will also be instructed to refrain from taking over the counter medications which may induce drowsiness throughout the duration of the study, and refrain from the use of any stimulants including caffeine for a minimum of 16 hours prior to study participation, avoid alcohol use for a minimum of 24 hours prior to participation, and avoid the use of nicotine for a minimum of 2 hours prior to the study. These are requested to obtain clean physiological recordings (e.g., Gilbert, Dibb, Plath, & Hiyane, 2000 [caffeine, nicotine]; Kähkӧnen, Wilenius, Nikulin, Ollikainen, & Ilmoniemi, 2003 [alcohol]). If the participant reports use of a stimulant, medication inducing drowsiness, nicotine, alcohol, or the actiwatch indicates less than 6 hours of rest, the participant will be released from the study for that day and asked to reschedule. In the event that the actiwatch fails, confirmation will rely on self-report and be recorded within the study log.

Following informed consent, subjects will complete a medical history questionnaire with a study physician that includes caffeine consumption habits to determine any possible side effects due to caffeine withdrawal. A member of the research team will measure and record the subject's vital signs (temperature, respiration rate, blood pressure, pulse, and oxygen saturation) on the medical history questionnaire. The study physician will review the medical history questionnaire and vital signs to make a final determination regarding eligibility. In addition to determining eligibility, the study physician or medical practitioner will discuss with the subject regular caffeine consumption habit and whether the subject is likely to experience any negative side effects associated with caffeine withdrawal (e.g., headache). If determined to be eligible by the study physician, subjects will then be enrolled in the study, complete the volunteer registry database form, receive the actiwatch and be provided verbal instructions on its use and be given a handout of participation guidelines. After receiving the actiwatch and guidelines, the subject will be offered the opportunity for stimulation familiarization. This will entail applying the stimulation at the prescribed intensity (2 mA) for a duration of 5 minutes, with the anode at F3 and cathode on the contralateral bicep (right arm). The purpose of this will be to allow the subject to experience what the stimulation feels like so that they know what to expect for the stimulation days. After stimulation has been applied, the electrodes will be removed and the subjects will complete the following questionnaires: demographic questionnaire, Morningness-Eveningness Questionnaire (MEQ) , Adult ADHD Self Report Scale (ASRS), Sleep Timing Questionnaire (STQ), Beck Depression Inventory (BDI), Shipley's Institute of Living Scale (SILS), Convergence Insufficiency Symptom Survey (CISS), Samn-Perelli Fatigue Scale, Short Stress State Questionnaire (SSSQ), Behavioral Inhibition / Avoidance Scales (BIS/BAS), Karolinska Sleepiness Scale (KSS), and Profile of Mood States - Short Form (POMS-SF). The subject will next complete a baseline session of the Rapid Visual Information Processing Task (RVIP) and Conners' Continuous Performance Task (CPT). Following completion of questionnaires, the electroencephalogram will be placed on the subjects and baseline measurements will be taken, which is a series of three computerized tasks provided by Advanced Brain Monitoring (ABM Tasks) which will be used for baseline, and pre- / post-stimulation EEG measurements. Subjects will then meet with the research pilot who will go over the flight tasks required of this study and escort the subject into the simulator for familiarization and baseline flight performance data collection. During the familiarization flight, the research pilot will ensure the subject is able to meet prescribed flight standards such as maintain specified headings, airspeeds and altitudes with minimal input/prompts, which will be recorded on the flight standards sheet. The baseline flight will consist of a scenario similar to, but not exact, as the scenarios that will be performed on treatment days. Baseline performance and EEG will be recorded and archived for analyses/interpretation. Subjects will be released at this point for the day.

Visits 2-3: tDCS stimulation test sessions.

Subjects will return for visit two at minimum 16 hours following their first visit. Visits two and three will be scheduled such that there is at least 48 hours in-between visits to avoid carry-over effects from stimulation application. Procedures for both visits will be the same. When the subject arrives, compliance with study instructions will be verified and recorded on the subject compliance sheet. If the subject does not comply with medication/stimulant/alcohol consumption instructions or the actiwatch indicates less than 6 hours of rest, the subject will be released from the study for that day and asked to reschedule. In the event that the actiwatch fails, confirmation will rely on self-report and be recorded in the study notebook.

Subjects will then complete the side effect questionnaire, KSS, Samn-Perelli Fatigue Scale, SSSQ and POMS-SF to determine whether any physical symptoms are present prior to stimulation (e.g., headaches) and any mood disturbances. Once questionnaires are completed, the subject's vital signs will be measured and recorded on the side effect questionnaire.

Next, the subject will be prepared for completing the flight scenarios and receiving stimulation. First, the subject will be fitted with the EEG and pre-stimulation baseline recordings will be obtained while the subject completes an additional iteration of the ABM tasks. Next, the scalp will be marked for tDCS electrode placement using a washable marker. This will be done as the EEG is removed so that the EEG electrode placements can be used to identify placement for tDCS electrodes. Scalp cleaning will occur as needed. Once removed, the subject will be escorted to the simulator where the tDCS electrodes will be put in place. The subject will be offered the opportunity to make adjustments as needed for comfort and to re-familiarize with the simulator. Once comfortable, a pre-flight mission brief will be given by the research pilot followed by the completion of a standard pre-flight checklist. These are estimated to last approximately 20 minutes total. Once the brief and checklist are completed, the flight scenario will begin. They have been designed to require minimal inputs by pilots and have been previously validated as low workload. Two flight scenarios were designed that include the same number of maneuvers, and require the same flight parameters (e.g., airspeed, altitude). One flight will involve a flight from Ft. Rucker to Montgomery and the other flight will be reversed (Montgomery to Ft. Rucker) so the subjects do not repeat the exact same flight twice. Thus, subjects will fly one scenario on visit two and a different one on visit three, which will be counterbalanced amongst subjects.

Timing of stimulation will differ by randomly assigning subjects to one of two groups. Group A will receive the active stimulation during the pre-mission brief and pre-flight checklist completion, for a total of 20 minutes, to evaluate whether application of stimulation at the start of the flight prevents the onset of degraded performance. Group B will receive the active stimulation at two time points, each for a duration of 10 minutes, for a total of 20 minutes. The first delivery of stimulation would occur at 30 minutes into the flight, while the second administration will occur at 60 minutes into the flight. This will be done to evaluate whether stimulation applied during the expected timeframe of loss of vigilance (approximately 30 minutes into the task) will offset this loss. To clarify, stimulus timing is a between-groups factor. A secondary task will also be implemented to measure whether performance changes occur on primary or secondary task performance. The secondary task will consist of periodic radio calls the pilot must respond to and physical responses to a visual targets presented on a tablet placed within the cockpit. Each group will also experience a sham-stimulation condition where at each of the intervals, stimulation will be applied for 10% of the stimulation period corresponding with their group assignments (Group A: 30s ramp up time, 60s stimulation, 30s ramp down time, for 2 minutes total; Group B: 2 deliveries with 30s ramp up time and 30s ramp down time, for 1 minute total).

At the completion of the flight the subject will be escorted out of the simulator, tDCS electrodes will be removed. The subject will complete the NASA TLX, side effect questionnaire, KSS, Samn-Perelli Fatigue Scale, SSQ, POMS-SF, and the BDI to determine whether any physical symptoms or sleepiness/mood changes may have occurred due to the stimulation. The physical side effect questionnaire and BDI will be examined immediately following completion to evaluate the score. If a score greater than five is obtained on the side effects questionnaire, the study physician will be notified and will consult with the subject to evaluate whether the reported symptoms are due to the stimulation and if the subject is safe to continue, needs to be rescheduled for another day, or needs to be removed from the study. After questionnaires have been completed, the EEG will be reapplied to record data while the participant completes one iteration of each the RVIP and CPT. Once all tasks are completed, the subject will complete a post-stimulation questionnaire (Appendix U) to evaluate whether the subject could detect differences between active and sham stimulation, and whether the subject thought the stimulation altered performance. Next, the subject will be escorted to the subject lounge. The subject will remain in the subject lounge where he will have access to activities (reading, TV, ping pong, etc.) for the next 8 hours. Every two hours after the first RVIP and CPT administration, another RVIP and CPT administration will be given, along with the physical side effect questionnaire, KSS, Samn-Perelli Fatigue Scale, SSSQ and POMS-SF. This will allow us to track the time course of the tDCS effects. After the final tasks and questionnaire administration, the subject will be released for the day and reminded to keep the actiwatch on to record any changes to sleep. As the third visit will be the final treatment visit, the participant will be requested to return the actiwatch at a time that is convenient, but at least 48 hours following the stimulation application to ensure measurement of at least two nights' sleep. Compensation will be contingent upon the return of the actiwatch device, as subjects will need to complete their 1099 tax form when returning the watch.

The total length of time for a test session is approximately twelve hours. Prior to release, a member of the research team will check vital signs, and then the subject will meet briefly with the study physician to determine whether the subject can safely be cleared and released for the day. Table 5 presents the time required for each activity. At the end of the third session the subject will be reminded to return the actiwatch in at least 48 hours and to continue wearing it until returning. Upon return of the actiwatch, the KSS will be administered once more. Finally, the post-study questionnaire will be administered to evaluate the usability/acceptance of tDCS.

ELIGIBILITY:
Inclusion Criteria:

1. Must be a male 18 (Active Duty) or 19 (National Guard, Reservist) to 40 years old.
2. Must be a rated rotary-wing aviator with at least 200 hours of total flight experience, and have flown (aircraft or simulator) within the past 6 months, assessed by self-report.
3. Must have a current DD-2292 (up-slip indicating clear for flight duties). Subjects will self-report this on the medical history questionnaire (Appendix A).
4. Must have obtained at minimum 6 hours of sleep prior to data collection, as assessed by actigraphy data and self-report.
5. Must have refrained from consumption of caffeine and medications that cause drowsiness, 16 hours, nicotine, 2 hours, and alcohol, 24 hours, prior to the study, assessed by self-report.

Exclusion Criteria:

1. Not having a current DD-2992.
2. The following medically-related exclusionary criteria will be used, as assessed and verified by the study physician (in addition to possessing a DD-2992):

   1. Currently taking medications which induce drowsiness, such as over-the-counter antihistamines. Any self-medication will be assessed through self-report
   2. No current medical conditions or medications affecting cognitive function or attention.
   3. Any history of any attention deficit condition requiring medication.
   4. Any history of psychological/psychiatric disorder.
   5. Any history of seizures, migraines, or neurological disorders.
   6. History of a head injury involving loss of consciousness.
   7. Any metal implanted within the head (e.g., shrapnel, surgical clips) or any implanted devices (e.g., cardiac pacemaker, brain stimulator, hydrocephalic shunt).
   8. Skin condition on the scalp, such as psoriasis or eczema, or wounds on the head.
   9. Currently receiving hormonal therapy treatments.
   10. Potential for caffeine withdrawal symptoms that will impede cognitive testing.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Rapid Visual Information Processing Task | 7 min
  Cognitive function - sustained attention The RVIP is a well-validated measure of sustained attention (Bakan, 1959). In each trial, subjects are presented with a sequence of digits and must detect "target" sequences within those presented. The target sequence is an even-odd-even string of numbers. When participants detect this string, they press the spacebar as quickly as possible. Difficulty is manipulated by changing the speed at which the numbers are presented (1 vs. 2 seconds).
Continuous Performance Task | 14 min
  Cognitive function - sustained attention The continuous performance task (Conners & Sitarenios, 2011) is a well validated measure of sustained attention and response inhibition. In this task, subjects are presented with a series of letters and are instructed to respond when they see any letter except for the letter X. Subjects are presented with 360 trials with varied intervals of 1, 2, and 4 seconds. Total time to complete this task is 14 minutes.
Flight performance - primary task | 90 min
  Simulated flight 90 min simulated flight scenario in a UH60 simulator.
Flight performance - secondary task | 90 min
  Simulated flight with visual secondary task A visual task presented during the flight requiring monitoring.
Response to emergency | 1 - 5 min
  Simulated emergency that requires response during flight.
Physiological response | 90 min
  EEG recording before and after stimulation.

SECONDARY OUTCOMES:
Flight experience | 10 min
  Demographic information
Behavioral Scales Behavioral Inhibition / Avoidance Scale | 10 min
  Trait Motivation The BIS/BAS scales are a valid and reliable set of scales that assess behavioral inhibition (BIS) and behavioral approach (BAS; Carver & White, 1994). The BAS provides three indices of behavioral approach: reward responsiveness (positive anticipation of rewarding events), drive (pursuit of rewards), and fun seeking (search for new rewarding situations). These scales provide a measurement of motivational behavioral systems.
Samn-Perelli Fatigue Scale | 1 min
  Fatigue The Samn-Perelli Fatigue Scale (Samn & Perelli, 1982) is a single item scale that has participants rate their current level of fatigue from 1 (fully alert, wide awake) to 7 (completely exhausted, unable to function effectively. The Samn-Perelli Fatigue Scale was included because it was initially developed to assess military aircrew fatigue and correlates with extended flight hours (r = .52, Samn & Perelli, 1982).
Short Stress State Questionnaire | 2 min
  Stress State The Short Stress State Questionnaire (Helton, 2004; Helton & Näswall, 2015) is a 24 item scale that measures the constructs of distress, worry, and task engagement. Each construct consists of eight items each.
40 Mini-Marker Personality Scale | 10 min
  This scale requires approximately 10 minutes to complete. Saucier (1994) developed a briefer version of a scale developed by Goldberg (1992) which uses 100 unipolar terms to describe personality traits based on the Big-Five Factor Structure (Tupes & Christal, 1992): agreeableness, conscientiousness, extraversion, neuroticism, and openness. The scale consists of 40 common human traits and subjects are were asked to rate how accurately these traits described themselves using a 9-point Likert scale.
Boredom Proneness Scale | 5 min
  The Boredom Proneness Scale is composed of 28 statements that participants rate on a scale from 1 (highly disagree) to 7 (highly agree). Reliability and validity of this instrument have been extensively studied and consistently shown to be strong (Vodanovich & Watt, 2016). This scale requires approximately 5 minutes to complete.

OTHER OUTCOMES:
Adult ADHD Self Report Scale Symptom Checklist | 2 min
  ADHD Symptoms The ASRS contains 18 items and requires 2 minutes for completion. It was developed in conjunction with the World Health Organization (WHO) and the Workgroup on Adult ADHD (Kessler et al., 2005) and is used as a screening tool with adult patients. The items are consistent with the Diagnostic and statistical manual of mental disorders, version IV criteria (American Psychiatric Association, 2000).
Sleep Timing Questionnaire | 3 min
  Sleep habits The STQ is an 18-item self-report measure of sleep habits and requires 3 minutes for completion. Research shows it to be valid (such that it correlates with sleep diary information) and reliable across repeated administrations (Monk et al., 2003).
Beck Depression Inventory | 2 min
  Depression symptoms Depression symptoms will be measured using the Beck Depression Inventory- II (BDI-II; Beck, Steer, & Brown, 1996). The BDI-II is a commonly used 21-item, multiple-choice self-report which captures affect, cognition, and physical symptoms of depression over the most recent two week period. Higher scores indicate greater endorsement of depression symptoms. It requires approximately 2 minutes to complete.
Karolinska Sleepiness Scale | 1 min
  Sleepiness The KSS is a well-validated single item questionnaire that asks subjects to rate how sleepy they feel at the moment (Kaida et al., 2006). The KSS measures daytime sleepiness with higher scores indicating greater daytime sleepiness. This requires approximately 1 minute to complete.
Convergence Insufficiency Symptom Survey | 2 min
  Convergence insufficiency The Convergence Insufficiency Symptom Survey (CISS; Borsting et al., 1999) is a 15-item questionnaire that ask participants to rate the severity of symptoms consistent with convergence insufficiency.
Shipley's Institute of Living Scale | 15 min
  Intelligence The SILS was designed to assess general intellectual functioning in adults and adolescents, and to aid in detecting cognitive impairment in individuals with normal original intelligence. The SILS yields three major summary scores: Vocabulary, Abstraction Quotient, and combined Total scores.
Profile of Mood States - Short Form | 3 min
  Mood symptoms The POMS-SF is a valid and reliable short version of the POMS, a measure of psychological distress and mood (McNair, Lorr, & Droppleman, 1981). The POMS-SF contains 35 items, in each an adjective is provided and the subject rates how much it describes them using a 5-point Likert scale format (Curran, Andrykowski, & Studts, 1995). It takes approximately 3 minutes to complete.
Symptom checklist | 2 min
  Side effects
Welch Allyn Connex 6000 | 5 min
  Physiology / health
NASA Task Load Index | 10 min
  Workload
Post Stimulation Questionnaire | 1 min
  Effects of stimulation
Post Study Questionnaire | 1 min
  Perceived usability of stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Katie Feltman, PhD, Principal Investigator — US Army Aeromedical Research Laboratory
Locations (1):
- U.S. Army Aeromedical Research Laboratory, Fort Rucker, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IDP.

DOCUMENTS (1):
  • Informed Consent Form (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/01/NCT04697901/ICF_000.pdf